CLINICAL TRIAL: NCT03244709
Title: Tocilizumab Dose-tapering and Interruption in Patients With Giant Cell Arteritis Achieving the Clinical Remission: a Prospective, Pilot Study.
Brief Title: Tocilizumab Dose-tapering and Interruption in Patients With Giant Cell Arteritis Achieving the Clinical Remission.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital of Prato (Other)
Responsible Party: Principal Investigator, Fabrizio Cantini, Director of the Dpt. of Rheumatology, Hospital of Prato
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Hospital of Prato, Italy
Record Dates: First submitted 2017-08-01; First posted 2017-08-09 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Giant Cell Arteritis
Keywords: Giant cell arteritis,; Tocilizumab; Aortitis; Remission
MeSH Terms: conditions — Giant Cell Arteritis; Aortitis | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with GCA (ACR 1990 criteria) (Experimental): At diagnosis, all GCA patients with or without involvement of aorta and its thoracic branches will receive PDN 50 mg/day and TCZ 8 mg/Kg/iv monthly. In all patients PDN dose will be reduced of 10 mg every 2 weeks until interruption at week 12.
  Week 12. Subcutaneous TCZ 162 mg/weekly will be administered for additional 12 weeks.
  Week 24. TCZ tapering every 8 weeks as follows:
  * 1 injection every 2 weeks
  * 1 injection every 3 weeks
  * 1 injection every 4 weeks Week 48. TCZ withdrawal. Week 72. Remission evaluation.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Intravenous Tocilizumab followed by subcutaneousTocilizumab

SUMMARY:
Interleukin-6 (IL-6), a pro-inflammatory cytokine, has been found to have a crucial role in the pathogenesis of Giant cel arteritis (GCA). Based on this rationale, several recent studies demonstrated the efficacy of tocilizumab (TCZ), an anti-IL-6 targeted monoclonal antibody, for the treatment of patients with refractory GCA. Confirming previous reports,in a recent retrospective study the investigators successfully treated 10 patient with refractory GCA with TCZ. All patients achieved a complete disease remission evaluated by clinical, laboratory, and positron emission tomography (PET). In a considerable number of GCA patients treated with corticosteroids (CS) the therapy may be interrupted with no disease flares. No data are available on the management of patients achieving the remission with TCZ.

DETAILED DESCRIPTION:
Study design. Open-label, prospective, pilot study on patients with giant cell arteritis (GCA) resistant to corticosteroids (CS) .

Setting. Rheumatology department, Hospital of Prato, Prato, Italy. Treatment. All refractory GCA patients with or without involvement of aorta and its thoracic branches treated with intravenous TCZ at the dose of 8 mg/Kg/monthly or subcutaneous TCZ at the dose of 162 mg/weekly who achieved a stable remission over a 6-month period should receive reduced TCZ doses with the following schedules: intravenous TCZ tapering to 2 mg/Kg/monthly with drug withdrawal at month 4, and subcutaneous TCZ monthly reduction through the lengthening of injection intervals every 2, 3 , and 4 weeks, and with drug interruption at month 4.

Primary end-point. To investigate the maintenance of clinical remission after TCZ interruption over a 6-month follow-up period.

Secondary end-points. To assess the maintenance of clinical remission during the treatment, to evaluate the role of acute-phase reactants and PET in predicting the relapse and remission, and to assess the occurrence of adverse event (AEs).

ELIGIBILITY:
Inclusion Criteria:

- All consecutive patients meeting the 1990 ACR classification criteria for GCA.

Exclusion Criteria:

* Corticosteroid treatment during the previous 6 months.
* Uncontrolled diabetes.
* Uncontrolled hypertension.
* History of cancer within the past 5 years.
* History of frequent infections in the past.
* Positivity of screening procedures for latent tuberculosis infection.
* Uncontrolled dyslipidemia at baseline.
* Known intestinal diverticulosis.
* Concomitant hematologic disorders.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients maintaining the off-therapy clinical remission over the follow-up as expressed by absence of GCA symptoms and signs, normal ESR and CRP values, absence of arterial wall inflammation at PET examination | 6-month off-therapy period
  ESR ≤15 mm/h; CRP ≤0.5 mg/dl; VAS pain ≤10; PET: normalized SUVmax ≤1

SECONDARY OUTCOMES:
The percentage of patients achieving and maintaining the clinical remission during the treatment with TCZ as expressed by the absence of GCA symptoms and signs, normal ESR and CRP values, absence of arterial wall inflammation at PET examination | 12 months
  Absence of GCA symptoms and signs, ESR ≤15 mm/h, CRP ≤0.5 mg/dL, PET: normalized SUVmax ≤1
To compare the role of acute-phase reactants and 18F-FDG-PET in the evaluation of remission. | Months 6,12,18
  Linear regression analysis for the correlation between ESR and CRP values and nSUVmax at baseline and after therapy
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0" MeDRA 12.1. | Month 18
  Overall AEs and serious AEs will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Fabrizio Cantini, Prato, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salvarani C, Cantini F, Hunder GG. Polymyalgia rheumatica and giant-cell arteritis. Lancet. 2008 Jul 19;372(9634):234-45. doi: 10.1016/S0140-6736(08)61077-6. PMID 18640460
- [Background] Soussan M, Nicolas P, Schramm C, Katsahian S, Pop G, Fain O, Mekinian A. Management of large-vessel vasculitis with FDG-PET: a systematic literature review and meta-analysis. Medicine (Baltimore). 2015 Apr;94(14):e622. doi: 10.1097/MD.0000000000000622. PMID 25860208
- [Background] Stone JH, Tuckwell K, Dimonaco S, Klearman M, Aringer M, Blockmans D, Brouwer E, Cid MC, Dasgupta B, Rech J, Salvarani C, Schett G, Schulze-Koops H, Spiera R, Unizony SH, Collinson N. Trial of Tocilizumab in Giant-Cell Arteritis. N Engl J Med. 2017 Jul 27;377(4):317-328. doi: 10.1056/NEJMoa1613849. PMID 28745999
- [Result] Unizony S, Arias-Urdaneta L, Miloslavsky E, Arvikar S, Khosroshahi A, Keroack B, Stone JR, Stone JH. Tocilizumab for the treatment of large-vessel vasculitis (giant cell arteritis, Takayasu arteritis) and polymyalgia rheumatica. Arthritis Care Res (Hoboken). 2012 Nov;64(11):1720-9. doi: 10.1002/acr.21750. PMID 22674883
- [Result] Loricera J, Blanco R, Hernandez JL, Castaneda S, Mera A, Perez-Pampin E, Peiro E, Humbria A, Calvo-Alen J, Aurrecoechea E, Narvaez J, Sanchez-Andrade A, Vela P, Diez E, Mata C, Lluch P, Moll C, Hernandez I, Calvo-Rio V, Ortiz-Sanjuan F, Gonzalez-Vela C, Pina T, Gonzalez-Gay MA. Tocilizumab in giant cell arteritis: Multicenter open-label study of 22 patients. Semin Arthritis Rheum. 2015 Jun;44(6):717-23. doi: 10.1016/j.semarthrit.2014.12.005. Epub 2014 Dec 27. PMID 25697557
- [Result] Proven A, Gabriel SE, Orces C, O'Fallon WM, Hunder GG. Glucocorticoid therapy in giant cell arteritis: duration and adverse outcomes. Arthritis Rheum. 2003 Oct 15;49(5):703-8. doi: 10.1002/art.11388. PMID 14558057